CLINICAL TRIAL: NCT02713776
Title: Reduction by Pasireotide of the Effluent Volume in High-output Enterostomy in Patients Refractory to Usual Medical Treatment : Phase II Multicentric Randomized Double Bland Placebo Controlled Study
Brief Title: Reduction by Pasireotide of the Effluent Volume in High-output Enterostomy in Patients Refractory to Usual Medical Treatment
Acronym: SOMILEO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014_880
Record Dates: First submitted 2016-02-29; First posted 2016-03-21 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Enterostomy
Keywords: High-Output Enterostomy; Pasireotide; Somatostatin Analogues
MeSH Terms: interventions — pasireotide

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Pasireotide (Experimental): Pasireotide 0.9 mg by subcutaneous injection twice a day during 3 days and 1 intramuscular injection of pasireotide Long Acting Release (LAR) 60mg on Day 4 morning.
  Interventions: Drug: Pasireotide
- Placebo (Placebo Comparator): Placebo by subcutaneous injection twice a day during 3 days and 1 intramuscular injection of placebo on Day 4 morning.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pasireotide — Pasireotide 0.9 mg by subcutaneous injection twice a day during 3 days and 1 intramuscular injection of pasireotide Long Acting Release (LAR) 60mg on Day 4 morning.
  Other Names: Pasireotide 0.9 mg (SIGNIFOR®) and Pasireotide 60mg Long Acting Release (LAR)
  Arms: Pasireotide
Drug: Placebo — Placebo by subcutaneous injection twice a day during 3 days and 1 intramuscular injection of placebo on Day 4 morning.
  Other Names: Placebo of pasireotide 0.9 mg by subcutaneous injection twice a day during 3 days and 1 intramuscular injection of pasireotide LAR (Long Acting Release) 60mg on Day 4
  Arms: Placebo

SUMMARY:
During rectal or complex digestive surgery with multiple digestive resections and anastomosis, the creation of enterostomy is a common procedure. In France, it is estimated that 20000 patients have an ileostomy and 16000 new digestive stomas are formed each year with approximately 30% of enterostomy. Enterostomy might sometimes give high-output not controlled with usual medical treatment (e.g loperamide ± codeine) and exposes the patients to important hydro-electrolytic loss leading to a risk for dehydration, electrolyte abnormalities and acute renal failure. This risk implies parenteral correction which may extend hospital stay and delay home return.

Somatostatin analogues (octreotide, lanreotide and pasireotide) could reduce digestive secretions and decrease digestive peristalsis. Nevertheless, somatostatin analogues are not routinely used for the treatment of patients with high-output enterostomy and their efficacy in the indication (off-label) was only tested in small case series. Pasireotide (SOM230, SIGNIFOR®) is currently indicated for the treatment of patients with Cushing's disease for whom surgery is not an option or for whom surgery has failed.

As the efficacity of pasireotide in patients with high-output enterostomy refractory to usual medical treatment associated with an oral fluid restriction has never been demonstrated before, there is a need to perform a pilot, double-blind, randomized, placebo-controlled trial evaluating its impact on reduction of the effluent volume.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female patients ≥ 18 years old ;
* Patients who underwent an intestinal surgery with enterostomy repair in the three weeks preceding the inclusion ;
* Patients with high-output ileostomy or jejunostomy > 1000 ml/24h ;
* Patients with failure of treatment combining oral fluid restriction and loperamide (up to 8 capsules/24h) +/- codeine syrup (10 mg x 3/24h) during 5 days ;
* Patients who gave its written informed consent to participate to the study ;
* Patients affiliated to a social insurance regime.

Exclusion Criteria:

* Male and Female patients < 18 years old ;
* Patients who did not give its written informed consent to participate to the study ;
* Patients who received somatostatin analogues during the month before inclusion ;
* Patients with symptomatic cholelithiasis or acute or chronic pancreatitis ;
* Patients with uncontrolled diabetes (with HbA1c (glycated hemoglobin) > 8%) ;
* Patients who are hypothyroid and not on adequate replacement therapy ;
* Patients who have congestive heart failure (NYHA (New York Heart Association) Class III or IV), unstable angina, sustained ventricular tachycardia, ventricular fibrillation, advanced heart block or a history of clinically significant bradycardia or acute myocardial infarction within the 6 months preceding randomization ;
* Patients with history of syncope or family history of idiopathic sudden death ;
* Patients with screening or baseline (predose) : QT interval corrected for heart rate using Fridericia's correction (QTcF) QTcF > 450 msec (male), QTcF > 460 msec (female) (QT interval corrected for heart rate using Fridericia's correction) ;
* Patients with not corrected hypokalaemia and/or hypomagnesaemia ;
* Patients with liver disease such as cirrhosis, chronic active hepatitis, or chronic persistent hepatitis, or patients with alanine transaminase/aspartate transaminase (ALT/AST) > 2 x Upper Limit of Normal (ULN), serum bilirubin > 2 x ULN ;
* Patients with Child-Pugh C cirrhosis ;
* Female patients who are pregnant or lactating, or are of childbearing potential and not practicing a medically acceptable method of birth control ;
* Patients with abnormal coagulation (PT and/or APTT elevated by 30% above normal limits) or patients receiving anticoagulants that affect PT (prothrombin time) or activated partial thromboplastin time (APTT) ;
* Patients with known hypersensitivity to somatostatin analogues or any other component of the pasireotide LAR ;
* Patients under guardianship ;
* Patients nonaffiliated to a social insurance regime.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2016-12-13 (Actual); Primary Completion 2021-01-08 (Actual); Study Completion 2021-01-08 (Actual)

PRIMARY OUTCOMES:
Compare the efficacy of pasireotide versus placebo in reduction of high-output | Evaluated 72 hours after first injection of treatment
  Decrease of enterostomy output (ml/24H)within the 72 hours after first injection of treatment

SECONDARY OUTCOMES:
Estimate the success rate of pasireotide and placebo | 1 week after first injection of treatment
  Number of normal renal function patients in both arms with an enterostomy output than 800 millimeters (mL) /24h within a week after first injection of treatment allowing discontinuation of intravenous perfusion.
Compare the decrease in the length of hospitalization with pasireotide versus placebo | 1 month after the end of treatment
  Duration of hospitalization in days in both arms
Compare the incidence of premature closure of stoma due to high-output with pasireotide versus placebo | 2 months after enterostomy creation
  Rate of premature closure of stoma due to high-output (before 2 months after creation) in both arms
Evaluate the economic impact of pasireotide in this indication | 2 months from the inclusion of the patient in the study
  Costs of taking care of patients from French Public Health Insurance perspective in both arms
Incidence of treatment - Emergent Adverse Events | during treatment (4 days), one week, two weeks, three weeks and one month after treatment
  Nature, number and grade of adverse events observed throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Eddy COTTE, Professor, Principal Investigator — Hospices Civils de Lyon - Centre Hospitalier Lyon Sud
Locations (14):
- France (14):
  - Chu Amiens-Picardie, Amiens
  - Chu Estaing, Clermont-Ferrand
  - Hopital Beaujon, Clichy
  - Chu Albert Michallon, La Tronche
  - Hôpital Claude HURIEZ - CHRU Lille, Lille
  - Centre Leon Berard, Lyon
  - Chu Marseille - Hopital Nord, Marseille
  - Institut Regional Du Cancer Val D'Aurelle, Montpellier
  - Chu Caremeau, Nîmes
  - Hopital Saint Antoine, Paris
  - Bordeaux Chu - Hopital Haut-Leveque, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Chu Rouen Ch. Nicolle, Rouen
  - Toulouse - Chu Purpan, Toulouse

REFERENCES:
- [Result] Beffara B, Hadj-Bouziane F, Hamed SB, Boehler CN, Chelazzi L, Santandrea E, Macaluso E. Dynamic causal interactions between occipital and parietal cortex explain how endogenous spatial attention and stimulus-driven salience jointly shape the distribution of processing priorities in 2D visual space. Neuroimage. 2022 Jul 15;255:119206. doi: 10.1016/j.neuroimage.2022.119206. Epub 2022 Apr 12. PMID 35427770